CLINICAL TRIAL: NCT01954264
Title: Epidemiology Study of Malariometric Determinants in Selected Post-Approval Programme Study Sites in Sub-Saharan Western Africa
Brief Title: Epidemiology Study of Malaria Transmission Intensity in Sub-Saharan Africa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 200187
Record Dates: First submitted 2013-09-19; First posted 2013-10-01 (Estimated); Results first posted 2018-10-05 (Actual); Last update posted 2020-01-21 (Actual); Status verified 2020-01

CONDITIONS: Malaria
Keywords: Saharan Western Africa; Epidemiology; Post-Approval Programme study; Malaria; Burden of Disease Study
MeSH Terms: conditions — Malaria | interventions — Data Collection

ARMS (1):
- Overall Study Group (Other): Subjects aged between 6 months to 9 years old, who were infected or not infected with Plasmodium falciparum parasite. Infection status was assessed using a blood smear slide and determined using microscopy.
  Interventions: Procedure: Capillary blood sample; Other: Data collection

INTERVENTIONS:
Procedure: Capillary blood sample — Capillary blood sample (up to 200µL) for determination of PP (blood slides).
Other: Data collection — Prospective data collection at the study visit by the internet based Electronic Case Report Form (eCRF)

SUMMARY:
This study is designed to characterise P. falciparum transmission intensity in subjects aged ≥6 months and <10 years by measurement of P. falciparum parasite prevalence, and to estimate the use of malaria control interventions at some centres selected for the EPI-MAL-002 and EPI-MAL-003 studies in sub-Saharan Western Africa.

DETAILED DESCRIPTION:
Two subsequent studies (EPI-MAL-002 and EPI-MAL-003) are planned to monitor vaccine safety prior to and after implementation of the RTS,S/AS01 candidate malaria vaccine. EPI-MAL-002 will take place before RTS,S is authorised and EPI-MAL-003 will start when RTS,S is registered and authorised in the country. A cross-sectional survey at peak transmission will provide by-site point estimates of Parasite prevalence (PP) and malaria control measure coverage in the areas participating in EPI-MAL-002/-003. EPI-MAL-006 will be conducted in advance of EPI-MAL-002/-003 in order to assess PP and malaria control measures to inform enrollment in these studies. The age group for enrollment (≥6 months - <10 years) will permit analysis of PP according to the World Health Organization (WHO) definition (2-9 years) and by the Joint Technical Expert Group (JTEG) suggested age (<5 years).

ELIGIBILITY:
Inclusion Criteria:

* Subjects' parent(s)/Legally Acceptable Representative(s) [LAR(s)] who, in the opinion of the investigator, can and will comply with the requirements of the protocol.
* A male or female equal or more than 6 months of age and less than 10 years of age at the time of survey.
* Signed informed consent or thumb-printed and witnessed informed consent obtained from the parent(s)/LAR(s) of the child.

Exclusion Criteria:

* Child in care.
* Current active participation in any trial involving administration of an investigational malaria vaccine or malaria drug.

Ages: 6 Months to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2421 (Actual)
Dates: Start 2013-10-19 (Actual); Primary Completion 2013-11-22 (Actual); Study Completion 2013-11-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (3):
- Burkina Faso (2):
  - GSK Investigational Site, Nouna
  - GSK Investigational Site, Ouagadougou
- GSK Investigational Site, Dakar, Senegal

IPD SHARING:
Plan to Share IPD: Yes
IPD is available via the Clinical Study Data Request site (click on the link provided below).
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below).
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com/Posting.aspx?ID=19801

REFERENCES:
- [Derived] Diallo A, Sie A, Sirima S, Sylla K, Ndiaye M, Bountogo M, Ouedraogo E, Tine R, Ndiaye A, Coulibaly B, Ouedraogo A, Faye B, Ba EH, Compaore G, Tiono A, Sokhna C, Ye M, Diarra A, Bahmanyar ER, De Boer M, Pircon JY, Usuf EA. An epidemiological study to assess Plasmodium falciparum parasite prevalence and malaria control measures in Burkina Faso and Senegal. Malar J. 2017 Feb 6;16(1):63. doi: 10.1186/s12936-017-1715-1. PMID 28166794
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — http://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: 200187 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 200187 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 200187 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 200187 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 200187 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 200187 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Overall Study Group
Started | 2421
Completed | 2421
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Overall Study Group
Number analyzed (Participants) | 2421
Age, Continuous [Mean (Standard Deviation); unit: Years] | 4.0 (2.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1155
  Male | 1266
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Plasmodium Falciparum (P. Falciparum) Parasitaemia (PFP), by Study Center
Description: PFP = measurement of parasite prevalence (PP) by center according to joint technical expert group (JTEG). Centers: Nouna-Burkina Faso (NOU-BF), Ouagadougou-Burkina Faso (OUA-BF), Keur Soce [Dakar area)-Senegal (DA-1-SE), Naikhar (Dakar area)-Senegal (DA-2-SE). A subject was defined as infected by P. falciparum parasitemia, if at least two of the subject's blood slide readings were positive for the corresponding parasitemia.
Time Frame: At Epoch 1 (Survey visit) (approximately 35 days)
Population: The According to Protocol (ATP) cohort included all evaluable subjects for whom at least one laboratory result of the blood sample was available.
Measure: Count of Participants; unit: Participants
Groups:
- 0.5-4Y Group: Subjects aged 6 months to 4 years (Y) old, who were infected or not infected with P. falciparum parasite. Infection status was assessed using a blood smear slide and determined using microscopy.
- 5-9Y Group: Subjects aged 5 to 9 years (Y) old, who were infected or not infected with P. falciparum parasite. Infection status was assessed using a blood smear slide and determined using microscopy.
Arm/Group | 0.5-4Y Group | 5-9Y Group
Number analyzed (Participants) | 1614 | 807
Participants
  NOU-BF: number analyzed (Participants) | 407 | 203
  NOU-BF | 235 | 153
  OUA-BF: number analyzed (Participants) | 399 | 201
  OUA-BF | 167 | 141
  DA-1-SE: number analyzed (Participants) | 399 | 204
  DA-1-SE | 2 | 1
  DA-2-SE: number analyzed (Participants) | 409 | 199
  DA-2-SE | 5 | 3
  Total | 409 | 298

2. Primary Outcome: Number of Subjects With Malaria Control Interventions (MCIs), Overall
Description: MCI = measurement of residual spraying, mosquito net usage, seasonal malaria chemoprevention (SMC), intermittent preventative treatment in infants (IPTi) and Artemisinin-based combination therapy (ACT) - therapy received within the last 14 days as indicator of malaria transmission intensity (MTI) by center and JTEG according to P. Falciparum infection status. Centers: Nouna-Burkina Faso (NOU-BF), Ouagadougou-Burkina Faso (OUA-BF), Keur Soce [Dakar area)-Senegal (DA-1-SE), Naikhar (Dakar area)-Senegal (DA-2-SE). Results presented for overall centers by the following characteristics: Use of Mosquito colis over 7 days (UMc > 7D), Use of Insecticide spray over 7 days (UIs > 7D), Use of Commercial Repellents over 7 days (UCR > 7D), Use of Traditional Repellents over 7 days (UTR > 7D), Use of none of above over 7 days (Una >7D), Use of indoor residual spray in past 12 months to spray interior walls (Uirs past 12M), Use of indoor residual spray - number of months ago (Uirs-nM)
Time Frame: At Epoch 1 (Survey visit) (approximately 35 days)
Population: The According to Protocol cohort included all evaluable subjects for whom at least one laboratory result of the blood sample was available.
Measure: Count of Participants; unit: Participants
Arm/Group | Overall Study Group
Number analyzed (Participants) | 2421
Participants
  UMc > 7D, Yes | 122
  UMc > 7D, Missing/No | 2299
  UIs > 7D, Yes | 65
  UIs > 7D, Missing/No | 2356
  UCR > 7D, Yes | 12
  UCR > 7D, Missing/No | 2409
  UTR > 7D, Yes | 278
  UTR > 7D, Missing/No | 2143
  Una >7D, Yes | 1979
  Una >7D, Missing/No | 442
  Uirs past 12M, Yes | 89
  Uirs past 12M, Missing/No | 2332
  Uirs-nM [1] | 0
  Uirs-nM [2] | 60
  Uirs-nM [3] | 8
  Uirs-nM [4] | 1
  Uirs-nM [5] | 0
  Uirs-nM [6] | 1
  Uirs-nM [7] | 0
  Uirs-nM [8] | 0
  Uirs-nM [9] | 18
  Uirs-nM [10] | 1
  Uirs-nM, Missing | 2332

3. Primary Outcome: Number of Subjects Infected With P.Falciparum Parasitemia Receiving Malaria Control Interventions (MCIs), by Infection Status
Description: as for outcome 2
Time Frame: At Epoch 1 (Survey visit) (approximately 35 days)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Groups:
- PF-INF Group: Subjects aged between 6 months to 9 years old, who were infected with P. falciparum parasite (PF-INF). Infection status was assessed using a blood smear slide and determined using microscopy.
- NOT-INF Group: Subjects aged between 6 months to 9 years old, who were not infected with P. falciparum parasite (NOT-INF). Infection status was assessed using a blood smear slide and determined using microscopy.
Arm/Group | PF-INF Group | NOT-INF Group
Number analyzed (Participants) | 707 | 1714
Participants
  Use of Mosquito coils over 7 days | 39 | 83
  Use of insecticide sprays over 7 days | 15 | 50
  Use of commercial repellents over 7 days | 4 | 8
  Use of traditional repellents over 7 days | 3 | 275
  Use of none of the above over 7 days | 649 | 1330
  Use of indoor residual spray in past 12 months | 3 | 86
  Use of indoor residual spray in past 1 month | 0 | 0
  Use of indoor residual spray in past 2 months | 1 | 59
  Use of indoor residual spray in past 3 months | 1 | 7
  Use of indoor residual spray in past 4 months | 0 | 1
  Use of indoor residual spray in past 5 months | 0 | 0
  Use of indoor residual spray in past 6 months | 1 | 0
  Use of indoor residual spray in past 7 months | 0 | 0
  Use of indoor residual spray in past 8 months | 0 | 0
  Use of indoor residual spray in past 9 months | 0 | 18
  Use of indoor residual spray in past 10 months | 0 | 1

4. Primary Outcome: Odds Ratio (OR) for the Number of Subjects With MCI, Infected With P. Falciparum Parasitemia, for the Nouna Center in Burkina Faso
Description: MCI = measurement of residual spraying, mosquito net usage, SMC, IPTi and ACT - therapy received within the last 14 days as indicator of MTI according to P. falciparum infection status. Note: - There was only the reference category available for 'Use of Traditional Repellents over 7 days': Missing/No - There was only one category available for 'Use of indoor residual spray - number of month ago': 2 Characteristics were as follows: Malaria treatment in past 14 days (Mt past 14D), Numbers of days of malaria treatment (NdMt), Other medication in the past 14 days (Om past 14D), Number of days of other medication (Ndom), Was the subject hospitalized in the last 3 months due to Malaria (Wsh3MM), Subject sleep under a mosquito net night before visit (Ssumnnbv), New net - less than 1 year (Nn < 1Y), Impregnated bednet (Ib), Pierced/torn bednet (P/tb), How many holes of that size (HS), UMc > 7D, UIs > 7D, UCR > 7D, UTR > 7D, Una >7D, Uirs past 12M.
Time Frame: At Epoch 1 (Survey visit) (approximately 35 days)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Unadjusted Odds Ratio
Arm/Group | PF-INF Group
Number analyzed (Participants) | 388
Unadjusted Odds Ratio
  MT PAST 14D, YES VS. NO | 0.323 [0.215 to 0.484]
  NDMT, ≥4 DAYS VS. ONGOING | 0.917 [0.051 to 16.494]
  NDMT, 1-3 DAYS VS. ONGOING | 0.596 [0.239 to 1.483]
  OM PAST 14D, YES VS. NO | 0.563 [0.403 to 0.788]
  NDOM, 1-7 DAYS VS. ONGOING | 1.155 [0.643 to 2.077]
  NDOM, ≥8 DAYS VS. ONGOING | NA [NA to NA] — Unadjusted OR value was not computable.
  WSH3MM, YES VS. NO | 0.612 [0.266 to 1.411]
  SSUMNNBV, YES VS. NO | 0.447 [0.165 to 1.216]
  NN < 1Y, YES VS. NO | 1.952 [0.742 to 5.138]
  IB, YES VS. NO | 0.677 [0.130 to 3.521]
  P/TB, YES VS. NO | 1.360 [0.550 to 3.359]
  HS, ≥5 VS. <5 | 0.311 [0.046 to 2.110]
  UMC > 7D, YES VS. MISSING/NO | 1.158 [0.631 to 2.125]
  UIS > 7D, YES VS. MISSING/NO | 0.456 [0.225 to 0.924]
  UCR > 7D, YES VS. MISSING/NO | 0.857 [0.142 to 5.169]
  UNA >7D, YES VS. MISSING/NO | 1.339 [0.840 to 2.134]
  UIRS PAST 12M, YES VS. NO | NA [NA to NA] — Unadjusted OR value was not computable.

5. Primary Outcome: Odds Ratio for the Number of Subjects With MCI, Infected With P. Falciparum Parasitemia, for the Ouagadougu Center in Burkina Faso
Description: MCI = measurement of residual spraying, mosquito net usage, SMC, IPTi and ACT - therapy received within the last 14 days as indicator of MTI according to P. falciparum infection status. Note: - There was only the reference category for 'Use of Insecticide spray over 7 days': Missing/No and 'Use of Traditional Repellents over 7 days': Missing/No - The reference category ('2') for 'Use of indoor residual spray - number of month ago': 2 Characteristics were as follows: Malaria treatment in past 14 days (Mt past 14D), Numbers of days of malaria treatment (NdMt), Other medication in the past 14 days (Om past 14D), Number of days of other medication (Ndom), Was the subject hospitalized in the last 3 months due to Malaria (Wsh3MM), Subject sleep under a mosquito net night before visit (Ssumnnbv), New net - less than 1 year (Nn < 1Y), Impregnated bednet (Ib), Pierced/torn bednet (P/tb), How many holes of that size (HS), UMc > 7D, UIs > 7D, UCR > 7D, UTR > 7D, Una >7D, Uirs past 12M.
Time Frame: At Epoch 1 (Survey visit) (approximately 35 days)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Unadjusted Odds Ratio
Arm/Group | PF-INF Group
Number analyzed (Participants) | 308
Unadjusted Odds Ratio
  MT PAST 14D, YES VS. NO | 0.143 [0.066 to 0.308]
  NDMT, ≥4 DAYS VS. ONGOING | NA [NA to NA] — Unadjusted OR value was not countable.
  NDMT, 1-3 DAYS VS. ONGOING | 0.341 [0.027 to 4.290]
  OM PAST 14D, YES VS. NO | 0.300 [0.171 to 0.529]
  NDOM, 1-7 DAYS VS. ONGOING | 0.568 [0.121 to 2.668]
  NDOM, ≥8 DAYS VS. ONGOING | NA [NA to NA] — Unadjusted OR value was not countable.
  WSH3MM, YES VS. NO | 1.146 [0.566 to 2.318]
  SSUMNNBV, YES VS. NO | 0.956 [0.510 to 1.791]
  NN < 1Y, YES VS. NO | 1.163 [0.486 to 2.785]
  IB, YES VS. NO | 0.699 [0.116 to 4.214]
  P/TB, YES VS. NO | 0.376 [0.072 to 1.956]
  HS, ≥5 VS. <5 | NA [NA to NA] — Unadjusted OR value was not countable.
  UMC > 7D, YES VS. MISSING/NO | 3.829 [0.425 to 34.458]
  UIS > 7D, YES VS. MISSING/NO | NA [NA to NA] — Unadjusted OR value was not countable.
  UCR > 7D, YES VS. MISSING/NO | NA [NA to NA] — Unadjusted OR value was not countable.
  UTR > 7D, NOT PERFORMED | NA [NA to NA] — Unadjusted OR value was not countable.
  UNA >7D, YES VS. MISSING/NO | 0.208 [0.024 to 1.793]
  UIRS PAST 12M, YES VS. NO | 0.948 [0.133 to 6.772]

6. Primary Outcome: Odds Ratio for the Number of Subjects With MCI, Infected With P. Falciparum Parasitemia, for the Keur Soce Center in Dakar Area in Senegal
Description: MCI = measurement of residual spraying, mosquito net usage, SMC, IPTi and ACT - therapy received within the last 14 days as indicator of MTI according to P. falciparum infection status. Note: - There was only one category available for 'Exact number of days of malaria treatment':1-3 days, 'Use of Indoor residual spray - numbers of months ago': 9, 'Use of Commercial Repellents over 7 days': Missing/No - There were not enough values in the reference category ('<5') to compute the OR for HS. Characteristics were as follows: Malaria treatment in past 14 days (Mt past 14D), Other medication in the past 14 days (Om past 14D), Number of days of other medication (Ndom), Was the subject hospitalized in the last 3 months due to Malaria (Wsh3MM), Subject sleep under a mosquito net night before visit (Ssumnnbv), New net - less than 1 year (Nn < 1Y), Impregnated bednet (Ib), Pierced/torn bednet (P/tb), UMc > 7D, UIs >7D, UCR > 7D, UTR > 7D, Una >7D.
Time Frame: At Epoch 1 (Survey visit) (approximately 35 days)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Unadjusted Odds Ratio
Arm/Group | PF-INF Group
Number analyzed (Participants) | 3
Unadjusted Odds Ratio
  MT PAST 14D, YES VS. NO | NA [NA to NA] — Unadjusted OR value was not computable.
  OM PAST 14D, YES VS. NO | 7.395 [0.656 to 83.396]
  NDOM, ≥ 8 days vs. Ongoing | NA [NA to NA] — Unadjusted OR value was not computable.
  NDOM, 1-7 days vs. Ongoing | NA [NA to NA] — Unadjusted OR value was not computable.
  WSH3MM, YES VS. NO | NA [NA to NA] — Unadjusted OR value was not computable.
  SSUMNNBV, YES VS. NO | 0.948 [0.085 to 10.523]
  NN < 1Y, YES VS. NO | NA [NA to NA] — Unadjusted OR value was not computable.
  IB, YES VS. NO | NA [NA to NA] — Unadjusted OR value was not computable.
  P/TB, YES VS. NO | NA [NA to NA] — Unadjusted OR value was not computable.
  UMC > 7D, YES VS. MISSING/NO | 5.383 [0.480 to 60.381]
  UIS > 7D, YES VS. MISSING/NO | NA [NA to NA] — Unadjusted OR value was not computable.
  UTR > 7D, YES VS. MISSING/NO | NA [NA to NA] — Unadjusted OR value was not computable.
  UNA >7D, YES VS. MISSING/NO | 0.484 [0.044 to 5.387]
  UIRS PAST 12M, YES VS. NO | NA [NA to NA] — Unadjusted OR value was not computable.

7. Primary Outcome: Odds Ratio for the Number of Subjects With MCI, Infected With P. Falciparum Parasitemia, for the Niakhar Center in Dakar Area in Senegal
Description: MCI = measurement of residual spraying, mosquito net usage, SMC, IPTi and ACT - therapy received within the last 14 days as indicator of MTI according to P. falciparum infection status. Note: - There was only one category available for 'Exact number of days of malaria treatment':1-3 days and 'How many holes of that size': ≥5. Characteristics were as follows: Malaria treatment in past 14 days (Mt past 14D), Numbers of days of malaria treatment (NdMt), Other medication in the past 14 days (Om past 14D), Number of days of other medication (Ndom), Was the subject hospitalized in the last 3 months due to Malaria (Wsh3MM), Subject sleep under a mosquito net night before visit (Ssumnnbv), New net - less than 1 year (Nn < 1Y), Impregnated bednet (Ib), Pierced/torn bednet (P/tb), How many holes of that size (HS), UMc > 7D, UIs > 7D, UCR > 7D, UTR > 7D, Una >7D, Uirs past 12M.
Time Frame: At Epoch 1 (Survey visit) (approximately 35 days)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Unadjusted Odds Ratio
Arm/Group | PF-INF Group
Number analyzed (Participants) | 8
Unadjusted Odds Ratio
  MT PAST 14D, YES VS. NO | NA [NA to NA] — Unadjusted OR value was not computable.
  OM PAST 14D, YES VS. N | 2.652 [0.525 to 13.404]
  NDOM, 1-7 DAYS VS. ONGOING | NA [NA to NA] — Unadjusted OR value was not computable.
  NDOM, ≥8 DAYS VS. ONGOING | 0.340 [0.020 to 5.764]
  WSH3MM, YES VS. NO | NA [NA to NA] — Unadjusted OR value was not computable.
  SSUMNNBV, YES VS. NO | NA [NA to NA] — Unadjusted OR value was not computable.
  NN < 1Y, YES VS. NO | NA [NA to NA] — Unadjusted OR value was not computable.
  IB, YES VS. NO | NA [NA to NA] — Unadjusted OR value was not computable.
  P/TB, YES VS. NO | 0.779 [0.184 to 3.299]
  UMC > 7D, YES VS. MISSING/NO | NA [NA to NA] — Unadjusted OR value was not computable.
  UIS > 7D, YES VS. MISSING/NO | NA [NA to NA] — Unadjusted OR value was not computable.
  UCR > 7D, YES VS. MISSING/NO | NA [NA to NA] — Unadjusted OR value was not computable.
  UTR > 7D, Yes vs. Missing/NO | 1.007 [0.238 to 4.255]
  UNA >7D, YES VS. MISSING/NO | 1.036 [0.245 to 4.375]
  UIRS PAST 12M, YES VS. NO | NA [NA to NA] — Unadjusted OR value was not computable.

8. Secondary Outcome: Number of Subjects With Other Medical History Characteristics, Overall
Description: The medical history characteristics were as follows: -subject sleep under a mosquito net night before visit (Ssumnnbv), New net - less than 1 year (Nn < 1Y), Impregnated Bednet (Ib), Pierced/torn bednet (P/tb), How many holes of that size (HS).
Time Frame: At Epoch 1 (Survey visit) (approximately 35 days)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Overall Study Group
Number analyzed (Participants) | 2421
Participants
  SSUMNNBV, YES | 2023
  SSUMNNBV, NO | 398
  NN < 1Y, YES | 1591
  NN < 1Y, NO | 431
  NN < 1Y, MISSING/NA | 399
  IB, YES | 1618
  IB, NO | 405
  IB, MISSING/NA | 398
  P/TB, YES | 406
  P/TB, NO | 1617
  P/TB, MISSING/NA | 398
  HS < 5 | 17
  HS ≥ 5 | 389
  HS, MISSING/NA | 2015

9. Secondary Outcome: Number of Subjects by Age, According to P. Falciparum Infection Status
Description: The annual age extended over a 0 year-9 years range. The age characteristics were summarized by P. falciparum infection status.
Time Frame: At Epoch 1 (Survey visit) (approximately 35 days)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Groups:
- PF-INF Group: Subjects aged between 6 months to 9 years (Y) old, who were infected with P. falciparum parasite (PF-INF). Infection status was assessed using a blood smear slide and determined using microscopy.
- NOT-INF Group: Subjects aged between 6 months to 9 years (Y) old, who were not infected with P. falciparum parasite (NOT-INF). Infection status was assessed using a blood smear slide and determined using microscopy.
Arm/Group | PF-INF Group | NOT-INF Group
Number analyzed (Participants) | 707 | 1714
Participants
  0 years olds | 48 | 202
  1 year olds | 98 | 380
  2 year olds | 131 | 348
  3 year olds | 71 | 136
  4 year olds | 61 | 139
  5 year olds | 55 | 106
  6 year olds | 53 | 109
  7 year olds | 59 | 104
  8 year olds | 66 | 92
  9 year olds | 65 | 98

10. Secondary Outcome: Number of Subjects by JTEG Age Group, According to P. Falciparum Infection Status
Description: The JTEG categorisation referred to the distribution of subjects by different age groups: 6 months to 4 years of age inclusive (0.5Y-4Y category) and 5 to 9 years of age inclusive (5-9Y category), tabulated according to P. falciparum infection status.
Time Frame: At Epoch 1 (Survey visit) (approximately 35 days)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | PF-INF Group | NOT-INF Group
Number analyzed (Participants) | 707 | 1714
Participants
  0.5Y - 4Y | 409 | 1205
  5Y - 9Y | 298 | 509

11. Secondary Outcome: Number of Subjects by Gender, According to P. Falciparum Infection Status
Description: The gender characteristics were summarized by P. falciparum infection status.
Time Frame: At Epoch 1 (Survey visit) (approximately 35 days)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | PF-INF Group | NOT-INF Group
Number analyzed (Participants) | 707 | 1714
Participants
  Female | 337 | 818
  Male | 370 | 896

12. Secondary Outcome: Number of Subjects With Plasmodium Species Other Than P. Falciparum, by JTEG Age Group and Per Total Centers
Description: Other Plasmodium species included: P. Malariae, P. Vivax, P. Ovale with Negative and Positive results. A subjects was defined as infected by a specified parasitemia if at least two of the subject's blood slide readings were positive for the corresponding parasitemia. The results were tabulated according to JTEG age categorisation.
Time Frame: At Epoch 1 (Survey visit) (approximately 35 days)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Groups:
- 0.5-4Y GROUP: Subjects aged between 6 months to 4 years (Y) old, who were infected or not infected with Plasmodium parasites. Infection status was assessed using a blood smear slide and determined using microscopy.
- 5-9Y GROUP: Subjects aged between 5 to 9 years (Y) old, who were infected or not infected with Plasmodium parasites. Infection status was assessed using a blood smear slide and determined using microscopy.
Arm/Group | 0.5-4Y GROUP | 5-9Y GROUP
Number analyzed (Participants) | 1614 | 807
Participants
  P. Malariae, Positive | 23 | 32
  P. Malariae, Negative | 1591 | 775
  P. Vivax, Positive | 0 | 0
  P. Vivax, Negative | 1614 | 807
  P. Ovale, Positive | 4 | 5
  P. Ovale, Negative | 1610 | 802

13. Secondary Outcome: Number of Subjects With Anti-malarial Therapy, Overall
Description: Anti-malarial therapy included Malaria treatment (MT) in past 14 days, Other medication (OM) in past 14 days and Malaria hospitalization (MH) in the last 3 months.
Time Frame: At Epoch 1 (Survey visit) (approximately 35 days)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Overall Study Group
Number analyzed (Participants) | 2421
Participants
  MT IN PAST 14 DAYS, YES | 187
  MT IN PAST 14 DAYS, NO | 2234
  OM IN PAST 14 DAYS, YES | 419
  OM IN PAST 14 DAYS, NO | 2002
  MH IN THE LAST 3 MONTHS, YES | 60
  MH IN THE LAST 3 MONTHS, NO | 2361

14. Secondary Outcome: Number of Days With Therapy, Overall
Description: The duration of anti-malarial therapy referred to the exact number of days of malaria treatment (EDMT) and the number of days of other medication (DOM). Note: * In case of several medication (malaria treatment or other medication) taken per subject, the maximum duration was computed for this study.
Time Frame: At Epoch 1 (Survey visit) (approximately 35 days)
Population: as for outcome 2
Measure: Number; unit: Days
Arm/Group | Overall Study Group
Number analyzed (Participants) | 2421
Days
  EDMT, Ongoing | 26
  EDMT, 1-3 days | 155
  EDMT, ≥ 4days | 3
  EDMT, Missing/NA | 2237
  DOM, Ongoing | 101
  DOM, 1-7 days | 310
  DOM, ≥ 8 days | 7
  DOM, Missing/NA | 2003

15. Secondary Outcome: Days of Malaria Treatment, Overall
Description: This endpoint presents results per total centers and across all age categories.
Time Frame: At Epoch 1 (Survey visit) (approximately 35 days)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Overall Study Group
Number analyzed (Participants) | 2421
Days | 3.0 (0.81)

16. Secondary Outcome: Number of Subjects With Fever, Overall
Description: Characteristics of fever were the following: Fever in the last 24 hours (F 24h) and Fever* at visit (F* at V). Note: *Fever set to Yes if temperature recorded at visit after axillary conversion was ≥ 37.5 ◦C.
Time Frame: At Epoch 1 (Survey visit) (approximately 35 days)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Overall Study Group
Number analyzed (Participants) | 2421
Participants
  F 24h, Yes | 331
  F 24h, No | 2090
  F* at V, Yes | 179
  F* at V, No | 2241
  F* at V, Missing | 1

17. Secondary Outcome: Days With Fever, Overall
Description: This endpoint presents results per total centers and across all age categories.
Time Frame: At Epoch 1 (Survey visit) (approximately 35 days)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Overall Study Group
Number analyzed (Participants) | 2421
Days | 3.0 (2.69)

18. Secondary Outcome: Number of Persons With P. Falciparum Living in the Same Part of the House of Persons Enrolled in the Study (PLSPH-PES), Overall
Description: The malaria prevention and risk factor presented in this endpoint was: Number of persons living in the same part of the house - persons enrolled in the study (PLSPH-PES), in the following combinations: < y/x, where x are persons enrolled in the study among less than y persons living in the same part of the house, y-z/x, where x are persons enrolled in the study among y to z persons living in the same part of the house, > z/x, where x persons are enrolled in the study among more than z persons living in the same part of the house, y-z/> x, where more than x persons enrolled in the study among y to z persons living in the same part of the house, > z/> x, where more than x persons enrolled in the study among more than z persons living in the same part of the house.
Time Frame: At Epoch 1 (Survey visit) (approximately 35 days)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Overall Study Group
Number analyzed (Participants) | 2421
Participants
  PLSPH-PES, <3/1 | 517
  PLSPH-PES, 4-5/1 | 590
  PLSPH-PES, >5/1 | 864
  PLSPH-PES, <3/2 | 54
  PLSPH-PES, 4-5/2 | 112
  PLSPH-PES, >5/2 | 214
  PLSPH-PES, <3/3 | 0
  PLSPH-PES, 4-5/3 | 15
  PLSPH-PES, >5/3 | 42
  PLSPH-PES, 4-5/>3 | 0
  PLSPH-PES, >5/>3 | 13

19. Secondary Outcome: Descriptive Statistics for Number of Persons With P. Falciparum Living in the Same Part of the House of Persons Enrolled in the Study (PLSPH-PES), Overall
Description: The malaria prevention and risk factor presented in this endpoint was: Number of persons living in the same part of the house (PLSPH).
Time Frame: At Epoch 1 (Survey visit) (approximately 35 days)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Persons Living in Same Part of House
Arm/Group | Overall Study Group
Number analyzed (Participants) | 2421
Persons Living in Same Part of House | 7.8 (6.49)

20. Secondary Outcome: Number of Subjects With Different P. Falciparum Parasite Densities, Living in the Same House, by Center
Description: The malaria prevention and risk factor for this endpoint was: Number of subjects living in the same part of the house - persons enrolled in the study (PLSPH-PES), in the following combinations: < y/x, where x are persons enrolled in the study among less than y persons living in the same part of the house, y-z/x, where x are persons enrolled in the study among y to z persons living in the same part of the house, > z/x, where x persons are enrolled in the study among more than z persons living in the same part of the house, y-z/> x, where more than x persons enrolled in the study among y to z persons living in the same part of the house, > z/> x, where more than x persons enrolled in the study among more than z persons living in the same part of the house. Results are presented for the Nouna-Burkina Faso (NOU-BF), Ouagadougou-Burkina Faso (OUA-BF), Keur Soce [Dakar area)-Senegal (DA-1-SE) and Naikhar (Dakar area)-Senegal (DA-2-SE) centers.
Time Frame: At Epoch 1 (Survey visit) (approximately 35 days)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Groups:
- Low PD Group: Subjects aged between 6 months to 9 years old, with low P. falciparum parasite density (<2500 parasite per µL).
- Medium PD Group: Subjects aged between 6 months to 9 years old, with medium P. falciparum parasite density (2500 - 9999 parasite per µL).
- High PD Group: Subjects aged between 6 months to 9 years old, with high P. falciparum parasite density (10000 - 19999 parasite per µL).
- Vhigh PD Group: Subjects aged between 6 months to 9 years old, with very high P. falciparum parasite density (≥20000 parasite per µL).
- Neg PD Group: Subjects aged between 6 months to 9 years old, who were not infected with P. falciparum parasite.
Arm/Group | Low PD Group | Medium PD Group | High PD Group | Vhigh PD Group | Neg PD Group
Number analyzed (Participants) | 411 | 164 | 70 | 62 | 1714
Participants
  NOU-BF, PLSP-PES, <3/1 | 85 | 34 | 14 | 11 | 68
  NOU-BF, PLSP-PES, 4-5/1 | 86 | 38 | 17 | 8 | 93
  NOU-BF, PLSP-PES, >5/1 | 49 | 22 | 6 | 4 | 57
  NOU-BF, PLSP-PES, <3/2 | 1 | 0 | 1 | 0 | 0
  NOU-BF, PLSP-PES, 4-5/2 | 4 | 2 | 2 | 0 | 4
  NOU-BF, PLSP-PES, >5/2 | 4 | 0 | 0 | 0 | 0
  NOU-BF, PLSP-PES, <3/3 | 0 | 0 | 0 | 0 | 0
  NOU-BF, PLSP-PES, 4-5/3 | 0 | 0 | 0 | 0 | 0
  NOU-BF, PLSP-PES, >5/3 | 0 | 0 | 0 | 0 | 0
  NOU-BF, PLSP-PES, 4-5/>3 | 0 | 0 | 0 | 0 | 0
  NOU-BF, PLSP-PES, >5/>3 | 0 | 0 | 0 | 0 | 0
  OUA-BF, PLSP-PES, <3/1 | 67 | 26 | 15 | 16 | 122
  OUA-BF, PLSP-PES, 4-5/1 | 44 | 24 | 12 | 14 | 100
  OUA-BF, PLSP-PES, >5/1 | 7 | 3 | 2 | 3 | 17
  OUA-BF, PLSP-PES, <3/2 | 16 | 3 | 0 | 1 | 24
  OUA-BF, PLSP-PES, 4-5/2 | 28 | 10 | 0 | 1 | 19
  OUA-BF, PLSP-PES, >5/2 | 5 | 1 | 0 | 1 | 7
  OUA-BF, PLSP-PES, <3/3 | 0 | 0 | 0 | 0 | 0
  OUA-BF, PLSP-PES, 4-5/3 | 7 | 0 | 0 | 1 | 1
  OUA-BF, PLSP-PES, >5/3 | 1 | 0 | 0 | 0 | 2
  OUA-BF, PLSP-PES, 4-5/>3 | 0 | 0 | 0 | 0 | 0
  OUA-BF, PLSP-PES, >5/>3 | 0 | 0 | 0 | 0 | 0
  DA-1-SE, PLSP-PES, <3/1 | 0 | 0 | 0 | 0 | 59
  DA-1-SE, PLSP-PES, 4-5/1 | 1 | 1 | 0 | 1 | 139
  DA-1-SE, PLSP-PES, >5/1 | 0 | 0 | 0 | 0 | 235
  DA-1-SE, PLSP-PES, <3/2 | 0 | 0 | 0 | 0 | 8
  DA-1-SE, PLSP-PES, 4-5/2 | 0 | 0 | 0 | 0 | 42
  DA-1-SE, PLSP-PES, >5/2 | 0 | 0 | 0 | 0 | 92
  DA-1-SE, PLSP-PES, <3/3 | 0 | 0 | 0 | 0 | 0
  DA-1-SE, PLSP-PES, 4-5/3 | 0 | 0 | 0 | 0 | 6
  DA-1-SE, PLSP-PES, >5/3 | 0 | 0 | 0 | 0 | 15
  DA-1-SE, PLSP-PES, 4-5/>3 | 0 | 0 | 0 | 0 | 0
  DA-1-SE, PLSP-PES, >5/>3 | 0 | 0 | 0 | 0 | 4
  DA-2-SE, PLSP-PES, <3/1 | 0 | 0 | 0 | 0 | 0
  DA-2-SE, PLSP-PES, 4-5/1 | 0 | 0 | 0 | 0 | 12
  DA-2-SE, PLSP-PES, >5/1 | 6 | 0 | 1 | 0 | 452
  DA-2-SE, PLSP-PES, <3/2 | 0 | 0 | 0 | 0 | 0
  DA-2-SE, PLSP-PES, 4-5/2 | 0 | 0 | 0 | 0 | 0
  DA-2-SE, PLSP-PES, >5/2 | 0 | 0 | 0 | 0 | 104
  DA-2-SE, PLSP-PES, <3/3 | 0 | 0 | 0 | 0 | 0
  DA-2-SE, PLSP-PES, 4-5/3 | 0 | 0 | 0 | 0 | 0
  DA-2-SE, PLSP-PES, >5/3 | 0 | 0 | 0 | 1 | 23
  DA-2-SE, PLSP-PES, 4-5/>3 | 0 | 0 | 0 | 0 | 0
  DA-2-SE, PLSP-PES, >5/>3 | 0 | 0 | 0 | 0 | 9

21. Secondary Outcome: Descriptive Statistics for Subjects With Different P. Falciparum Parasite Densities, Living in the Same House, by Center
Description: The malaria prevention and risk factor for this endpoint was: Number of subjects living in the same part of the house (PLSPH). Results are presented for the Nouna-Burkina Faso (NOU-BF), Ouagadougou-Burkina Faso (OUA-BF), Keur Soce [Dakar area)-Senegal (DA-1-SE) and Naikhar (Dakar area)-Senegal (DA-2-SE) centers.
Time Frame: At Epoch 1 (Survey visit) (approximately 35 days)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Persons Living in Same Part of House
Arm/Group | Low PD Group | Medium PD Group | High PD Group | Vhigh PD Group | Neg PD Group
Number analyzed (Participants) | 411 | 164 | 70 | 62 | 1714
Persons Living in Same Part of House
  NOU-BF, PLSPH | 4.5 (2.29) | 4.6 (2.48) | 4.2 (1.30) | 4.2 (1.68) | 4.7 (2.21)
  OUA-BF, PLSPH | 3.8 (1.21) | 3.8 (1.20) | 3.7 (1.14) | 3.7 (1.45) | 3.8 (1.23)
  DA-1-SE, PLSPH | 5.0 (0.00) | 5.0 (0.00) | NA (NA) — No results were available with the specified criteria. | 4.0 (0.00) | 8.0 (4.94)
  DA-2-SE, PLSPH | 16.2 (5.91) | NA (NA) — No results were available with the specified criteria. | 9.0 (0.00) | 9.0 (0.00) | 15.0 (7.73)

22. Secondary Outcome: Number of Subjects With P. Falciparum by Situation Area, Overall
Description: The malaria prevention and risk factor characteristics for this endpoint were the following: Situation area (rural, urban, semi-rural) and Type of Location*. Note: *Large city = >1 million habitants; Small city = >50000 & < 1 million habitants ; Town = > 10000 and < 50000 habitants; Countryside = < 10000 habitants.
Time Frame: At Epoch 1 (Survey visit) (approximately 35 days)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Overall Study Group
Number analyzed (Participants) | 2421
Participants
  Situation area, Rural | 2127
  Situation area, Urban | 294
  Situation area, Semi-rural | 0
  Type of Location, Large city | 14
  Type of Location, Small city | 0
  Type of Location, Town | 282
  Type of Location, Countryside | 2125

23. Secondary Outcome: Number of Subjects With Different P. Falciparum Densities by Situation Area and Center
Description: The malaria prevention and risk factor characteristics were the following: Situation area (urban, rural, semi-rural) and Type of Location*. Note: *Large city = >1 million habitants; Small city = >50000 & < 1 million habitants ; Town = > 10000 and < 50000 habitants; Countryside = < 10000 habitants. Results are presented for the Nouna-Burkina Faso (NOU-BF), Ouagadougou-Burkina Faso (OUA-BF), Keur Soce [Dakar area)-Senegal (DA-1-SE) and Naikhar (Dakar area)-Senegal (DA-2-SE) centers.
Time Frame: At Epoch 1 (Survey visit) (approximately 35 days)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Low PD Group | Medium PD Group | High PD Group | Vhigh PD Group | Neg PD Group
Number analyzed (Participants) | 411 | 164 | 70 | 62 | 1714
Participants
  NOU-BF, Situation area, Rural | 129 | 71 | 23 | 16 | 84
  NOU-BF, Situation area, Urban | 100 | 25 | 17 | 7 | 138
  NOU-BF, Situation area, semi-rural | 0 | 0 | 0 | 0 | 0
  NOU-BF, Type of Location, Large city | 0 | 1 | 0 | 0 | 0
  NOU-BF, Type of Location, Small city | 0 | 0 | 0 | 0 | 0
  NOU-BF, Type of Location, Town | 97 | 25 | 16 | 7 | 135
  NOU-BF, Type of Location, Countryside | 132 | 70 | 24 | 16 | 87
  OUA-BF, Situation area, Rural | 174 | 67 | 27 | 37 | 289
  OUA-BF, Situation area, Urban | 1 | 0 | 2 | 0 | 3
  OUA-BF, Situation area, semi-rural | 0 | 0 | 0 | 0 | 0
  OUA-BF, Type of Location, Large city | 2 | 0 | 1 | 0 | 5
  OUA-BF, Type of Location, Small city | 0 | 0 | 0 | 0 | 0
  OUA-BF, Type of Location, Town | 0 | 0 | 0 | 0 | 0
  OUA-BF, Type of Location, Countryside | 173 | 67 | 28 | 37 | 287
  DA-1-SE, Situation area, Rural | 1 | 1 | 0 | 1 | 600
  DA-1-SE, Situation area, Urban | 0 | 0 | 0 | 0 | 0
  DA-1-SE, Situation area, semi-rural | 0 | 0 | 0 | 0 | 0
  DA-1-SE, Type of Location, Large city | 0 | 0 | 0 | 0 | 5
  DA-1-SE, Type of Location, Small city | 0 | 0 | 0 | 0 | 0
  DA-1-SE, Type of Location, Town | 0 | 0 | 0 | 0 | 0
  DA-1-SE, Type of Location, Countryside | 1 | 1 | 0 | 1 | 595
  DA-2-SE, Situation area, Rural | 6 | 0 | 1 | 1 | 599
  DA-2-SE, Situation area, Urban | 0 | 0 | 0 | 0 | 1
  DA-2-SE, Situation area, semi-rural | 0 | 0 | 0 | 0 | 0
  DA-2-SE, Type of Location, Large city | 0 | 0 | 0 | 0 | 0
  DA-2-SE, Type of Location, Small city | 0 | 0 | 0 | 0 | 0
  DA-2-SE, Type of Location, Town | 0 | 0 | 0 | 0 | 2
  DA-2-SE, Type of Location, Countryside | 6 | 0 | 1 | 1 | 598

24. Secondary Outcome: Number of Subjects With P. Falciparum by House Construction Material and Other House Information, Overall
Description: The malaria prevention and risk factor characteristics for this endpoint were the following: - Main house construction material (MHCM) walls, floor, roof, windows/eaves, nets; - Main source of drinking water (MSDW); - Presence of electricity (PE). Note: *Natural floor = earth, sand, dung; Rudimentary floor = wood planks, palm, bamboo. % Closed water source (piper water, tube well, dug well, protected well); Open water source (unprotected well, spring water, rainwater, tanker truck, surface water).
Time Frame: At Epoch 1 (Survey visit) (approximately 35 days)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Overall Study Group
Number analyzed (Participants) | 2421
Participants
  MHCM walls, mud | 1176
  MHCM walls, brick | 728
  MHCM walls, cement/plaster | 140
  MHCM walls, cement/paint | 365
  MHCM walls, other | 12
  MHCM floor, natural floor* | 1283
  MHCM floor, rudimentary floor* | 16
  MHCM floor, vinyl oe asphalt strips | 95
  MHCM floor, ceramic tiles | 43
  MHCM floor, cement | 980
  MHCM floor, carpet | 3
  MHCM floor, other | 1
  MHCM roof, glass/palm | 632
  MHCM roof, iron sheet | 1493
  MHCM roof, tiles | 290
  MHCM roof, missing | 6
  MHCM windows/eaves, closed | 968
  MHCM windows/eaves, open | 653
  MHCM windows/eaves, partially open | 405
  MHCM windows/eaves, missing | 395
  MHCM nets, not present | 2005
  MHCM nets, present on all windows | 16
  MHCM nets, present on some windows | 6
  MHCM nets, missing | 394
  MSDW, bottled water | 2
  MSDW, closed water source % | 1706
  MSDW, open water source % | 712
  MSDW, not applicable | 1
  PE, Yes | 361
  PE, No | 2060

25. Secondary Outcome: Number of Subjects With Different P. Falciparum Parasite Densities, by House Information and Center
Description: The malaria prevention and risk factor characteristics for this endpoint were the following: - Main house construction material (MHCM) walls, floor, roof, windows/eaves, nets; - Main source of drinking water (MSDW); - Presence of electricity (PE). Natural floor = earth, sand, dung; Rudimentary floor = wood planks, palm, bamboo. Closed water source = pipe water, tube well, dug well, protected well; Open water source = unprotected well, spring water, rainwater, tanker truck, surface water. Results are presented for the Nouna-Burkina Faso (NOU-BF), Ouagadougou-Burkina Faso (OUA-BF), Keur Soce [Dakar area)-Senegal (DA-1-SE) and Naikhar (Dakar area)-Senegal (DA-2-SE) centers.
Time Frame: At Epoch 1 (Survey visit) (approximately 35 days)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Low PD Group | Medium PD Group | High PD Group | Vhigh PD Group | Neg PD Group
Number analyzed (Participants) | 411 | 164 | 70 | 62 | 1714
Participants
  MHCM walls, mud : NOU-BF | 49 | 18 | 4 | 6 | 52
  MHCM walls, mud : OUA-BF | 174 | 67 | 29 | 37 | 283
  MHCM walls, mud : DA-1-SE | 1 | 1 | 0 | 1 | 170
  MHCM walls, mud : DA-2-SE | 4 | 0 | 1 | 0 | 279
  MHCM walls, brick : NOU-BF | 153 | 70 | 32 | 17 | 129
  MHCM walls, brick : OUA-BF | 1 | 0 | 0 | 0 | 6
  MHCM walls, brick : DA-1-SE | 0 | 0 | 0 | 0 | 210
  MHCM walls, brick : DA-2-SE | 0 | 0 | 0 | 0 | 110
  MHCM walls, cement/plaster : NOU-BF | 6 | 1 | 1 | 0 | 12
  MHCM walls, cement/plaster : OUA-BF | 0 | 0 | 0 | 0 | 3
  MHCM walls, cement/plaster : DA-1-SE | 0 | 0 | 0 | 0 | 0
  MHCM walls, cement/plaster : DA-2-SE | 2 | 0 | 0 | 0 | 114
  MHCM walls, cement/paint : NOU-BF | 21 | 5 | 3 | 0 | 29
  MHCM walls, cement/paint : OUA-BF | 0 | 0 | 0 | 0 | 0
  MHCM walls, cement/paint : DA-1-SE | 0 | 0 | 0 | 0 | 220
  MHCM walls, cement/paint : DA-2-SE | 0 | 0 | 0 | 0 | 87
  MHCM walls, other : NOU-BF | 0 | 2 | 0 | 0 | 0
  MHCM walls, other : OUA-BF | 0 | 0 | 0 | 0 | 0
  MHCM walls, other : DA-1-SE | 0 | 0 | 0 | 0 | 0
  MHCM walls, other : DA-2-SE | 0 | 0 | 0 | 0 | 10
  MHCM floor, natural floor : NOU-BF | 114 | 66 | 17 | 11 | 90
  MHCM floor, natural floor : OUA-BF | 156 | 57 | 25 | 32 | 255
  MHCM floor, natural floor : DA-1-SE | 1 | 1 | 0 | 1 | 118
  MHCM floor, natural floor : DA-2-SE | 0 | 0 | 1 | 1 | 332
  MHCM floor, rudimentary floor : NOU-BF | 0 | 0 | 0 | 0 | 0
  MHCM floor, rudimentary floor : OUA-BF | 0 | 0 | 0 | 0 | 0
  MHCM floor, rudimentary floor : DA-1-SE | 0 | 0 | 0 | 0 | 0
  MHCM floor, rudimentary floor : DA-2-SE | 0 | 0 | 0 | 0 | 16
  MHCM floor, vinyl or asphalt strips : NOU-BF | 0 | 0 | 0 | 0 | 0
  MHCM floor, vinyl or asphalt strips : OUA-BF | 0 | 0 | 0 | 0 | 0
  MHCM floor, vinyl or asphalt strips : DA-1-SE | 0 | 0 | 0 | 0 | 95
  MHCM floor, vinyl or asphalt strips : DA-2-SE | 0 | 0 | 0 | 0 | 0
  MHCM floor, ceramic tiles : NOU-BF | 1 | 0 | 0 | 0 | 3
  MHCM floor, ceramic tiles : OUA-BF | 0 | 0 | 0 | 0 | 0
  MHCM floor, ceramic tiles : DA-1-SE | 0 | 0 | 0 | 0 | 36
  MHCM floor, ceramic tiles : DA-2-SE | 0 | 0 | 0 | 0 | 3
  MHCM floor, cement : NOU-BF | 114 | 30 | 23 | 12 | 129
  MHCM floor, cement : OUA-BF | 19 | 10 | 4 | 5 | 37
  MHCM floor, cement : DA-1-SE | 0 | 0 | 0 | 0 | 349
  MHCM floor, cement : DA-2-SE | 1 | 0 | 0 | 0 | 247
  MHCM floor, carpet : NOU-BF | 0 | 0 | 0 | 0 | 0
  MHCM floor, carpet : OUA-BF | 0 | 0 | 0 | 0 | 0
  MHCM floor, carpet : DA-1-SE | 0 | 0 | 0 | 0 | 2
  MHCM floor, carpet : DA-2-SE | 0 | 0 | 0 | 0 | 1
  MHCM floor, other : NOU-BF | 0 | 0 | 0 | 0 | 0
  MHCM floor, other : OUA-BF | 0 | 0 | 0 | 0 | 0
  MHCM floor, other : DA-1-SE | 0 | 0 | 0 | 0 | 0
  MHCM floor, other : DA-2-SE | 0 | 0 | 0 | 0 | 1
  MHCM roof, glass/palm : NOU-BF | 5 | 5 | 0 | 0 | 5
  MHCM roof, glass/palm : OUA-BF | 52 | 27 | 9 | 12 | 68
  MHCM roof, glass/palm : DA-1-SE | 1 | 1 | 0 | 1 | 100
  MHCM roof, glass/palm : DA-2-SE | 4 | 0 | 1 | 1 | 300
  MHCM roof, iron sheet : NOU-BF | 121 | 34 | 21 | 7 | 128
  MHCM roof, iron sheet : OUA-BF | 123 | 40 | 20 | 25 | 224
  MHCM roof, iron sheet : DA-1-SE | 0 | 0 | 0 | 0 | 451
  MHCM roof, iron sheet : DA-2-SE | 2 | 0 | 0 | 0 | 297
  MHCM roof, tiles : NOU-BF | 103 | 57 | 19 | 16 | 89
  MHCM roof, tiles : OUA-BF | 0 | 0 | 0 | 0 | 0
  MHCM roof, tiles : DA-1-SE | 0 | 0 | 0 | 0 | 3
  MHCM roof, tiles : DA-2-SE | 0 | 0 | 0 | 0 | 3
  MHCM windows/eaves, closed : NOU-BF | 79 | 26 | 16 | 5 | 84
  MHCM windows/eaves, closed : OUA-BF | 80 | 32 | 17 | 15 | 116
  MHCM windows/eaves, closed : DA-1-SE | 0 | 0 | 0 | 0 | 28
  MHCM windows/eaves, closed : DA-2-SE | 5 | 0 | 1 | 1 | 463
  MHCM windows/eaves, open : NOU-BF | 102 | 47 | 10 | 12 | 87
  MHCM windows/eaves, open : OUA-BF | 49 | 12 | 6 | 13 | 90
  MHCM windows/eaves, open : DA-1-SE | 0 | 0 | 0 | 0 | 88
  MHCM windows/eaves, open : DA-2-SE | 1 | 0 | 0 | 0 | 136
  MHCM windows/eaves, partially open : NOU-BF | 48 | 23 | 14 | 6 | 51
  MHCM windows/eaves, partially open : OUA-BF | 46 | 23 | 6 | 9 | 86
  MHCM windows/eaves, partially open : DA-1-SE | 0 | 0 | 0 | 0 | 92
  MHCM windows/eaves, partially open : DA-2-SE | 0 | 0 | 0 | 0 | 1
  MHCM nets, not present : NOU-BF | 224 | 95 | 40 | 23 | 215
  MHCM nets, not present : OUA-BF | 173 | 66 | 29 | 37 | 291
  MHCM nets, not present : DA-1-SE | 0 | 0 | 0 | 0 | 206
  MHCM nets, not present : DA-2-SE | 6 | 0 | 1 | 1 | 598
  MHCM nets, present on all windows : NOU-BF | 4 | 1 | 0 | 0 | 5
  MHCM nets, present on all windows : OUA-BF | 1 | 1 | 0 | 0 | 0
  MHCM nets, present on all windows : DA-1-SE | 0 | 0 | 0 | 0 | 2
  MHCM nets, present on all windows : DA-2-SE | 0 | 0 | 0 | 0 | 2
  MHCM nets, present on some windows : NOU-BF | 1 | 0 | 0 | 0 | 2
  MHCM nets, present on some windows : OUA-BF | 1 | 0 | 0 | 0 | 1
  MHCM nets, present on some windows : DA-1-SE | 0 | 0 | 0 | 0 | 1
  MHCM nets, present on some windows : DA-2-SE | 0 | 0 | 0 | 0 | 0
  MSDW, bottled water : NOU-BF | 0 | 0 | 0 | 0 | 0
  MSDW, bottled water : OUA-BF | 1 | 0 | 0 | 0 | 1
  MSDW, bottled water : DA-1-SE | 0 | 0 | 0 | 0 | 0
  MSDW, bottled water : DA-2-SE | 0 | 0 | 0 | 0 | 0
  MSDW, closed water source : NOU-BF | 146 | 57 | 24 | 9 | 116
  MSDW, closed water source : OUA-BF | 152 | 50 | 25 | 31 | 247
  MSDW, closed water source : DA-1-SE | 1 | 0 | 0 | 1 | 465
  MSDW, closed water source : DA-2-SE | 2 | 0 | 0 | 1 | 379
  MSDW, open water source : NOU-BF | 83 | 39 | 16 | 14 | 105
  MSDW, open water source : OUA-BF | 22 | 17 | 4 | 6 | 44
  MSDW, open water source : DA-1-SE | 0 | 1 | 0 | 0 | 135
  MSDW, open water source : DA-2-SE | 4 | 0 | 1 | 0 | 221
  MSDW, not applicable : NOU-BF | 0 | 0 | 0 | 0 | 1
  MSDW, not applicable : OUA-BF | 0 | 0 | 0 | 0 | 0
  MSDW, not applicable : DA-1-SE | 0 | 0 | 0 | 0 | 0
  MSDW, not applicable : DA-2-SE | 0 | 0 | 0 | 0 | 0
  PE, Yes : NOU-BF | 46 | 11 | 7 | 3 | 76
  PE, Yes : OUA-BF | 0 | 0 | 0 | 0 | 0
  PE, Yes : DA-1-SE | 0 | 0 | 0 | 0 | 164
  PE, Yes : DA-2-SE | 0 | 0 | 0 | 0 | 0
  PE, No : NOU-BF | 183 | 85 | 33 | 20 | 146
  PE, No : OUA-BF | 175 | 67 | 29 | 37 | 292
  PE, No : DA-1-SE | 1 | 1 | 0 | 1 | 436
  PE, No : DA-2-SE | 6 | 0 | 1 | 1 | 546

ADVERSE EVENTS:
Description: As planned per protocol, other (non-serious) adverse events were not collected.
Arm/Group | Overall Study Group
All-Cause Mortality (participants affected / at risk) | 0/2421
Serious Adverse Events (participants affected / at risk) | 0/2421
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.